CLINICAL TRIAL: NCT01578889
Title: A Phase 1 Trial to Evaluate the Safety, Tolerability, and Immunogenicity of an IL-12 pDNA Enhanced HIV-1 Multiantigen pDNA Vaccine Delivered Intramuscularly With Electroporation, With an HIV-1 rVSV Vaccine Boost, in Healthy HIV-Uninfected Adult Participants
Brief Title: Evaluating the Safety of and Immune Response to HIV-MAG DNA Vaccine With or Without Plasmid IL-12 Adjuvant Delivered Intramuscularly Via Electroporation Followed by VSV-gag HIV Vaccine Boost in Healthy, HIV-Uninfected Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 087; 11673 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Electroporation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Group 1: Vaccine (Experimental): At study entry and Months 1 and 3, participants will receive HIV-MAG vaccine administered as 0.5 mL by intramuscular (IM) injection in both the left and right deltoids using the Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device. At Month 6, they will receive the VSV HIV gag vaccine by IM injection in both the left and right deltoids.
  Interventions: Biological: HIV-MAG vaccine; Biological: VSV HIV gag vaccine; Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device
- Group 1: Placebo (Placebo Comparator): At study entry and Months 1 and 3, participants will receive placebo administered as 0.5 mL by IM injection in both the left and right deltoids using the Ichor Medical Systems TDS EP device. At Month 6, they will receive placebo by IM injection in both the left and right deltoids.
  Interventions: Biological: Placebo; Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device
- Group 2: Vaccine (Experimental): At study entry and Months 1 and 3, participants will receive HIV-MAG vaccine admixed with 250 mcg IL-12 pDNA adjuvant, and divided into two 0.55 mL IM injections administered in both the left and right deltoids using the Ichor Medical Systems TDS EP device. At Month 6, they will receive the VSV HIV gag vaccine by IM injection in both the left and right deltoids.
  Interventions: Biological: HIV-MAG vaccine; Biological: IL-12 pDNA adjuvant; Biological: VSV HIV gag vaccine; Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device
- Group 2: Placebo (Placebo Comparator): At study entry and Months 1 and 3, participants will receive placebo administered as 0.55 mL by IM injection in both the left and right deltoids using the Ichor Medical Systems TDS EP device. At Month 6, they will receive placebo by IM injection in both the left and right deltoids.
  Interventions: Biological: Placebo; Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device
- Group 3: Vaccine (Experimental): At study entry and Months 1 and 3, participants will receive HIV-MAG vaccine admixed with 1,000 mcg of the IL-12 pDNA adjuvant and divided into two 0.75 mL IM injections administered in both the left and right deltoids using the Ichor Medical Systems TDS EP device. At Month 6, they will receive the VSV HIV gag vaccine by IM injection in both the left and right deltoids.
  Interventions: Biological: HIV-MAG vaccine; Biological: IL-12 pDNA adjuvant; Biological: VSV HIV gag vaccine; Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device
- Group 3: Placebo (Placebo Comparator): At study entry and Months 1 and 3, participants will receive placebo administered as 0.75 mL by IM injection in both the left and right deltoids using the Ichor Medical Systems TDS EP device. At Month 6, they will receive placebo by IM injection in both the left and right deltoids.
  Interventions: Biological: Placebo; Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device
- Group 4: Vaccine (Experimental): At study entry and Months 1 and 3, participants will receive HIV-MAG vaccine admixed with 1500 mcg of the IL-12 pDNA adjuvant divided into two 0.9 mL IM injections administered in both the left and right deltoids using the Ichor Medical Systems TDS EP device. At Month 6, they will receive the VSV HIV gag vaccine by IM injection in both the left and right deltoids.
  Interventions: Biological: HIV-MAG vaccine; Biological: IL-12 pDNA adjuvant; Biological: VSV HIV gag vaccine; Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device
- Group 4: Placebo (Placebo Comparator): At study entry and Months 1 and 3, participants will receive placebo administered as 0.9 mL by IM injection in both the left and right deltoids using the Ichor Medical Systems TDS EP device. At Month 6, they will receive placebo by IM injection in both the left and right deltoids.
  Interventions: Biological: Placebo; Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device

INTERVENTIONS:
Biological: HIV-MAG vaccine — Participants assigned to receive the HIV-MAG vaccine will receive 3 mg of the vaccine with bupivacaine, alone or admixed with one of three doses of the IL-12 pDNA adjuvant.
  Arms: Group 1: Vaccine; Group 2: Vaccine; Group 3: Vaccine; Group 4: Vaccine
Biological: IL-12 pDNA adjuvant — Participants assigned to receive the IL-12 plasmid (IL-12 pDNA) adjuvant will receive one of three doses (total of 250 mcg, 1000 mcg, or 1500 mcg) of the adjuvant admixed with the HIV-MAG vaccine.
  Arms: Group 2: Vaccine; Group 3: Vaccine; Group 4: Vaccine
Biological: VSV HIV gag vaccine — Participants assigned to receive the VSV HIV gag vaccine will receive a total dose of 1x10^8 plaque-forming units (PFUs) administered as 5x10^7 PFU in 1 mL by IM injection in both the left and right deltoids at Month 6.
  Arms: Group 1: Vaccine; Group 2: Vaccine; Group 3: Vaccine; Group 4: Vaccine
Biological: Placebo — Placebo will consist of sodium chloride for injection, USP 0.9%.
  Arms: Group 1: Placebo; Group 2: Placebo; Group 3: Placebo; Group 4: Placebo
Device: Ichor Medical Systems TriGrid™ Delivery System (TDS) electroporation (EP) device — The HIV-MAG vaccine, IL-12 pDNA adjuvant, and placebos for IL-12 pDNA adjuvant/HIV-MAG vaccines will be delivered IM into the deltoid by the Ichor Medical Systems TDS EP device.

SUMMARY:
Some vaccines may work better when given together with another substance known as an adjuvant or when given with an experimental procedure called electroporation (EP). EP is a method where an electric pulse is administered to the same muscle where the vaccine injection is given. The addition of the adjuvant to the vaccine and the delivery with EP may increase a person's immune response to the vaccine. Combination approaches such as a DNA vaccine followed by live vector boost may also increase a person's immune response to the vaccine components. All of these interventions will be tested in this study.

This study will evaluate the safety and tolerability of and immune response to an HIV DNA vaccine with or without plasmid IL-12 adjuvant, when given by EP and followed by a live vector vaccine given IM by needle and syringe in healthy, HIV-uninfected adults.

DETAILED DESCRIPTION:
The effectiveness of a vaccine may be increased when combined with an adjuvant and/or when given with EP. The addition of an adjuvant or EP may increase a person's immune response to a vaccine. Furthermore, the immune response to HIV antigens may be improved by giving a DNA vaccine boosted with a live vector vaccine. The purpose of this study is to evaluate the safety, tolerability, and immunogenicity of an HIV DNA vaccine (HIV-MAG) alone or in combination with an IL-12 pDNA adjuvant, delivered IM via EP followed by a Vesicular Stomatitis Virus (VSV) HIV gag vaccine boost given IM by needle and syringe in healthy, HIV-uninfected adults.

Participants will be enrolled into the study in one of four groups. Each of the four groups will receive 3 mg of the HIV-MAG vaccine alone or combined with one of three different doses of the IL-12 pDNA adjuvant, followed by the VSV HIV gag vaccine boost. Within each of the four groups, participants will be randomly assigned to receive the study vaccines or placebo. At study entry (Day 0), all participants will undergo a physical examination and blood collection. Female participants will also take a pregnancy test. Participants will complete questionnaires and receive counseling on HIV risk reduction. They will also receive their first vaccination. Participants will remain in the clinic for 30 minutes after the vaccination for observation and monitoring.

Additional vaccination study visits will occur at Months 1, 3, and 6. At Months 1 and 3, participants will receive the same vaccine or placebo they received at study entry; at Month 6, participants will receive the VSV HIV gag vaccine or placebo. For 3 days after the study entry and Months 1 and 3 vaccination visits, participants will record their symptoms in a diary. After the Month 6 vaccination visit, participants will record their symptoms for 7 days.

Participants in Groups 1 and 3 will attend additional study visits on Days 1, 3, 14, 42, 91, 98, 169, 171, 175, 182, 273, and 364. Participants in Groups 2 and 4 will attend additional study visits on Days 14, 42, 98, 182, 273, and 364. Most study visits will include a physical examination, blood collection, oral mucosa examination, interviews and questionnaires, and oral mucosa examination. If participant has any oral sores, oral swabs may be collected. Saliva also may be collected. Select study visits will include a mini mental state exam, urine collection, HIV testing, and risk reduction counseling. Study researchers will contact participants at Months 15, 24, and 36 for follow-up health monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willing to be followed for the planned duration of the study
* Able and willing to provide informed consent
* Assessment of understanding: participant demonstrates understanding of this study and completes a questionnaire prior to the first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Willing to receive HIV test results
* Willing to discuss HIV infection risks, amenable to HIV risk reduction counseling, and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
* Willing to be contacted annually after completion of scheduled clinic visits for a total of 3 years following initial study injection
* Agrees not to enroll in another study of an investigational research agent prior to completion of last required protocol clinic visit (excludes annual contacts for safety surveillance)
* In good general health as shown by medical history, physical exam, and screening laboratory tests
* Assessed by the clinic staff as being at "low risk" for HIV infection
* Hemoglobin greater than or equal to 11.0 g/dL for participants who were born female; greater than or equal to 13.0 g/dL for participants who were born male
* White blood cell (WBC) count equal to 3,300 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 125,000 to 550,000/mm^3
* Chemistry panel: ALT, AST, alkaline phosphatase, and creatinine values less than or equal to the institutional upper limits of normal; CPK less than or equal to 2.0 times the institutional upper limit of normal
* Negative HIV-1 and -2 blood test: participants in the United States must have a negative Food and Drug Administration (FDA)-approved immunoassay
* Negative hepatitis B surface antigen (HBsAg)
* Negative anti-hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive
* Normal urine:

  1. Negative urine glucose, and
  2. Negative or trace urine protein, and
  3. Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis within institutional normal range)
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to vaccination on the day of initial vaccination
* Reproductive status: A participant who was born female must agree to consistently use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit; or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation; or be sexually abstinent. More information on this criterion can be found in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

* Allergy to amide-type local anesthetics (bupivacaine [Marcaine], lidocaine [Xylocaine], mepivacaine [Polocaine/Carbocaine], etidocaine [Duranest], prilocaine [Citanest, EMLA® cream])
* Presence of implanted electronic medical device (e.g., pacemaker, implantable cardioverter defibrillator)
* Presence of surgical or traumatic metal implant in the upper limb and/or upper torso
* Sinus bradycardia (defined as less than 50 bpm on exam) or a history of cardiac arrhythmia: e.g., supraventricular tachycardia, atrial fibrillation, or frequent ectopy
* Neurological or neuropsychiatric disorder that may interfere with the assessment of safety: e.g., frequent recurring headaches (i.e., a pattern of more than one headache per month affecting activities of daily living [ADLs]/work, frequent or severe/complicated migraines, cluster headaches), a chronic pain syndrome, dizziness, history of meningitis or encephalitis, cranial/spinal/peripheral neuropathy, limb weakness or paralysis, movement disorder, narcolepsy, stroke with sequelae, moderate/severe major depressive disorder, moderate/severe bipolar disorder
* Seizure disorder
* Untreated or incompletely treated syphilis infection
* HIV vaccine(s) received in a prior HIV vaccine trial. For potential participants who have received control/placebo in an HIV vaccine trial, the HVTN 087 Protocol Safety Review Team (PSRT) will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made for vaccines that have subsequently undergone licensure by the FDA. For potential participants who have received control/placebo in an experimental vaccine trial, the HVTN 087 PSRT will determine eligibility on a case-by-case basis. For potential participants who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the PSRT on a case-by-case basis.
* Immunosuppressive medications received within 168 days before first vaccination. (Not excluded: [1] corticosteroid nasal spray for allergic rhinitis; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids given for non-chronic conditions not expected to recur [length of therapy 10 days or less with completion at least 30 days prior to enrollment].)
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 60 days before first vaccination
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection (e.g., measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Investigational research agents received within 30 days before first vaccination
* Intent to participate in another study of an investigational research agent during the planned duration of the HVTN 087 study
* Influenza vaccine or any vaccines that are not live attenuated vaccines and were received within 14 days prior to first vaccination (e.g., tetanus, pneumococcal, hepatitis A or B)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. More information on this criterion can be found in the protocol.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent
* Serious adverse reactions to vaccines, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded: a participant who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Autoimmune disease
* Immunodeficiency
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the protocol.
* Diabetes mellitus type 1 or type 2, including cases controlled with diet alone. (Not excluded: history of isolated gestational diabetes.)
* Thyroidectomy, or thyroid disease requiring medication during the last 12 months
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema
* Hypertension:

  1. If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these participants, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  2. If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Body mass index (BMI) greater than or equal to 40; or BMI greater than or equal to 35 with two or more of the following: age greater than 45 years old, systolic blood pressure greater than 140 mm Hg, diastolic blood pressure greater than 90 mm Hg, current smoker, or known hyperlipidemia
* Deltoid skin fold measurement by caliper greater than 40 mm
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, platelet disorder requiring special precautions)
* Cancer (Not excluded: a participant with a surgical excision and subsequent observation period that in the investigator's estimation has a reasonable assurance of sustained cure or is unlikely to recur during the period of the study.)
* Asplenia: any condition resulting in the absence of a functional spleen
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are people with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of local injection/EP site reactogenicity signs and symptoms | Measured through Month 12
  Pain, tenderness, erythema, induration, and maximum severity of pain and/or tenderness
Frequency and severity of systemic reactogenicity signs and symptoms | Measured through Month 12
  Fever, malaise/fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and maximum severity of systemic symptoms
Magnitude of local injection/EP site pain as measured by a visual analog scale | Measured through Month 12
Frequency of adverse events (AEs) categorized by MedDRA body system, MedDRA preferred term, severity, and assessed relationship to study products | Measured through Month 12
  Detailed description of all AEs meeting DAIDS criteria for expedited reporting
Distribution of values of safety laboratory measures | Measured through Month 12
  White blood cells, neutrophils, lymphocytes, hemoglobin, alkaline phosphatase, platelets, alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine, and creatine phosphokinase (CPK) at baseline and at follow-up visits postvaccination
Number of participants with early discontinuation of vaccinations and reason for discontinuation | Measured through Month 12
Distribution of responses to questions regarding acceptability of study injections procedures | Measured through Month 12

SECONDARY OUTCOMES:
Response rate of CD4 T-cell responses measured by intracellular cytokine staining (ICS) for IFN-γ and/or IL-2, to HIV potential T-cell epitope (PTE) peptide pools representing Gag, Pol, Env, Nef, Tat, and Vif | Measured through Month 12
Response rate of CD8 T-cell responses measured by ICS for IFN-γ and/or IL-2, to HIV PTE peptide pools representing Gag, Pol, Env, Nef, Tat, and Vif | Measured through Month 12
Response rate of T-cell responses as measured by IFN-γ enzyme-linked immunospot (ELISpot) | Measured through Month 12
Induction of binding antibodies to HIV-1 gag p55 and HIV-1 6101 env gp160 | Measured through Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Christine (Mhorag) Hay, Study Chair — University of Rochester
Locations (5):
- United States (5):
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee

REFERENCES:
- [Background] Egan MA, Megati S, Roopchand V, Garcia-Hand D, Luckay A, Chong SY, Rosati M, Sackitey S, Weiner DB, Felber BK, Pavlakis GN, Israel ZR, Eldridge JH, Sidhu MK. Rational design of a plasmid DNA vaccine capable of eliciting cell-mediated immune responses to multiple HIV antigens in mice. Vaccine. 2006 May 22;24(21):4510-23. doi: 10.1016/j.vaccine.2005.08.024. Epub 2005 Aug 19. PMID 16140439
- [Background] Dolter KE, Evans CF, Ellefsen B, Song J, Boente-Carrera M, Vittorino R, Rosenberg TJ, Hannaman D, Vasan S. Immunogenicity, safety, biodistribution and persistence of ADVAX, a prophylactic DNA vaccine for HIV-1, delivered by in vivo electroporation. Vaccine. 2011 Jan 17;29(4):795-803. doi: 10.1016/j.vaccine.2010.11.011. Epub 2010 Nov 19. PMID 21094270
- [Background] Hirao LA, Wu L, Khan AS, Hokey DA, Yan J, Dai A, Betts MR, Draghia-Akli R, Weiner DB. Combined effects of IL-12 and electroporation enhances the potency of DNA vaccination in macaques. Vaccine. 2008 Jun 13;26(25):3112-20. doi: 10.1016/j.vaccine.2008.02.036. Epub 2008 Mar 11. PMID 18430495
- [Background] Johnson JE, Coleman JW, Kalyan NK, Calderon P, Wright KJ, Obregon J, Ogin-Wilson E, Natuk RJ, Clarke DK, Udem SA, Cooper D, Hendry RM. In vivo biodistribution of a highly attenuated recombinant vesicular stomatitis virus expressing HIV-1 Gag following intramuscular, intranasal, or intravenous inoculation. Vaccine. 2009 May 14;27(22):2930-9. doi: 10.1016/j.vaccine.2009.03.006. Epub 2009 Mar 13. PMID 19428903
- [Derived] Elizaga ML, Li SS, Kochar NK, Wilson GJ, Allen MA, Tieu HVN, Frank I, Sobieszczyk ME, Cohen KW, Sanchez B, Latham TE, Clarke DK, Egan MA, Eldridge JH, Hannaman D, Xu R, Ota-Setlik A, McElrath MJ, Hay CM; NIAID HIV Vaccine Trials Network (HVTN) 087 Study Team. Safety and tolerability of HIV-1 multiantigen pDNA vaccine given with IL-12 plasmid DNA via electroporation, boosted with a recombinant vesicular stomatitis virus HIV Gag vaccine in healthy volunteers in a randomized, controlled clinical trial. PLoS One. 2018 Sep 20;13(9):e0202753. doi: 10.1371/journal.pone.0202753. eCollection 2018. PMID 30235286
- [Derived] Li SS, Kochar NK, Elizaga M, Hay CM, Wilson GJ, Cohen KW, De Rosa SC, Xu R, Ota-Setlik A, Morris D, Finak G, Allen M, Tieu HV, Frank I, Sobieszczyk ME, Hannaman D, Gottardo R, Gilbert PB, Tomaras GD, Corey L, Clarke DK, Egan MA, Eldridge JH, McElrath MJ, Frahm N; NIAID HIV Vaccine Trials Network. DNA Priming Increases Frequency of T-Cell Responses to a Vesicular Stomatitis Virus HIV Vaccine with Specific Enhancement of CD8+ T-Cell Responses by Interleukin-12 Plasmid DNA. Clin Vaccine Immunol. 2017 Nov 6;24(11):e00263-17. doi: 10.1128/CVI.00263-17. Print 2017 Nov. PMID 28931520